CLINICAL TRIAL: NCT05888935
Title: Detection of Periapical Lesions on Dental Panoramic Images Based on Artificial Intelligence Using Cone Beam Computed Tomography
Brief Title: Detection of Periapical Lesions on Dental Panoramic Radiographs Based on Artificial Intelligence
Acronym: OPTITOMO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-04Obs-CHRMT
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Periapical Diseases
Keywords: tomography; dental injury; artificial intelligence; periapical lesions
MeSH Terms: conditions — Periapical Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dental periapical damages can have various reasons and is reflected by a radiolucent lesion on complementary imaging: angulated retro-alveolar (RA) radiographs, dental panoramic radiographs, and three-dimensional imaging such as computed tomography (CT) or cone-beam computed tomography (CBCT).

For the radiographic detection of these deep periodontal lesions, the dental panoramic represents a first approach commonly performed with relatively low radiation. The investigation can be followed by retroalveolar radiology imaging that are more localized and more precise. However, using these techniques, the detection rates of these lesions are low (20% and 36% respectively), it is necessary to use three-dimensional tomographic investigation to be more discriminating (69%). The gold standard imaging for detection of these lesions is CBCT followed by retroalveolar radiography (~2x less sensitive than CBCT) and panoramic radiography (~2x less sensitive than RA). Although not a full-thickness radiograph, the dental panoramic has the advantage of being more commonly performed while being less radiating than CBCT and giving a global view of the dental arches on a single image.

The detection of periapical lesions is done after a clinical assessment and a visual appreciation of the complementary examinations.

The aim of this project is to improve the detection of periapical lesions, by developing an algorithm able to identify them on a panoramic dental radiograph. This algorithm is based on a deep learning system trained with reference data including panoramic dental imaging and CBCT with an acquisition interval of less than 3 months. The model is based on a previous work, will improve the quality of the initial data (using CBCT), using innovative artificial intelligence algorithms (transfer learning).

DETAILED DESCRIPTION:
The final objective of the research is to improve the early diagnosis of periapical lesions, which would allow a better and faster care of these lesions namely at early stages. This represents a major public health interest since these lesions can be responsible for multiple local and regional pathologies (osteomyelitis, cervico-facial cellulitis, thrombophlebitis, cerebral abscesses...) or even more serious general pathologies (cardiac pathologies, cardiovascular diseases, diabetes, renal diseases, tendinopathies...). For certain target groups such as the military and high-level athletes, this research would make it possible to improve the assessment carried out before medical aptitude or club transfer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had CBCT and panoramic dental imaging with less than 3 months between the two examinations

Exclusion Criteria:

* Patients who refused to participe in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with periapical lesions
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Artificial Intelligence software performance | 2 years
  measurement of the F1 score. The F1 score is calculated as the harmonic mean of the precision and recall scores.
  It ranges from 0-100%, and a higher F1 score denotes a better quality classifier.

SECONDARY OUTCOMES:
Artificial Intelligence software specificity | 2 years
  measurement of the true positives, true negatives, false positives, false negatives

CONTACTS AND LOCATIONS:
Overall Officials: Marc ENGELS-DEUTSCH, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy; Paul RETIF, MD, PhD, Study Chair — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No